CLINICAL TRIAL: NCT01988597
Title: Dry Eye Symptoms and Quality of Life
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Senior Consultant, Singapore National Eye Centre
Other Study IDs: R1047/62/2013; 2013/595/A (Other: SingHealth Centralised Institutional Review Board)
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Dry Eyes
Keywords: Dry Eyes; Quality of life; Utility assessment
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dry Eyes
  Interventions: Other: Dry eyes

INTERVENTIONS:
Other: Dry eyes

SUMMARY:
Dry eye syndrome is a very common condition with multiple etiologies that includes systemic and ocular disease that causes reduction in the production of tears, as well as increase in tears evaporation. As a result of the various etiologies and large variability of dry eye's clinical sign, it has been a challenge for practitioners to have a consistent system to classify dry eyes and to have an appropriate and accurate measurement to quantify the severity of dry eyes and its impact on patients' quality of life.6 To date, no study which evaluates the extent of questionnaires correlates with changes in quality of life. With this cross sectional interview study, we aim to determine the efficacy of the questionnaires as a practical tool in our future clinical trials at our center.

DETAILED DESCRIPTION:
Dry eye is a multifactorial condition that affects 5-35% of the population.1 Common symptoms of this condition include eye irritation, heaviness of the eyelids, visual disturbances, tearing and light sensitivity.2 This condition significantly decrease patient health related quality of life (HRQOL). Clinical studies shown poor correlation between clinical test symptoms and self perceived severity of the disease.7 Studies also have shown that utilities of more severe dry eye similar to condition such as class III/IV angina affecting the QOL.6 Correlation between reduce quality of life and presenting symptoms is unknown compared to other factors such as cost and inconvenience of treatment. This implicates on the management of the condition. In addition, there is a significant socioeconomic burden. In 2009, 54,051 patients sought treatment for dry eye in the Singapore National Eye Centre (SNEC). In total, the costs for dry eye medication amounted to $181,354.17.4

Although different questionnaires have been used in assessment of dry eye, to date, there has been no study which evaluates the extent of questionnaires correlate with change in quality of life.

This is particularly important since symptoms of dry eyes are episodic and questionnaires administered at one time point may or may not reflect the true disease morbidity. Two of such questionnaires are the SPEED questionnaires which consist of 2 questions graded on a scale of 0-3 on frequency and grade 0-4 on severity and SANDE questionnaires which consist of 3 questions based on symptoms of frequency and severity.

Both of the questionnaires have been published and validated and utilized in the eye clinic by the investigators.

Over the last few years, SNEC/SERI has built up a dedicated team of dry eye researchers for trials and evaluation of diagnostic devices. There is an increasing interest internationally, especially from industry, to partner us for testing of commercial products.

Clinical importance Dry eye is a common and growing public health problem with significant morbidity and decrease in health related quality of life. Uncertainty in correlation between decrease quality of life with presenting symptoms and factors such as cost and inconvenience of treatment may implicate the management of the disease. For instance, if presenting symptoms correlate poorly with the perceived quality of life, more emphasis should be placed on making treatment more accessible and convenient. If there is a high correlation, the focus should be making current treatments more efficacious to relieve presenting symptoms.

The findings of this study will help us to decide the efficacy of the questionnaires use in future clinical trials in our centre.

Study Objectives and Purpose

1. To determine if the symptoms of dry eye assessed by the SPEED questionnaire correlate with utility values (HRQOL)
2. To determine if the symptoms of dry eye assessed by the SANDE questionnaire correlate with utility values (HRQOL)
3. To evaluate if the extent of correlation with HRQOL differs significantly between SPEED and SANDE questionnaires

   Study design:

   Prospective cross-sectional interview study

   Rationale Dry eye disease defined by The National Eye Institute Workshop as tear deficiency and excessive tear evaporation that causes damage to the ocular surface and is associated with symptoms and ocular discomfort.5 These symptoms causes adverse effect on quality of life (HRQL) of patients resulting in inappropriate management. In order to achieve a better correlation between dry eye symptoms and quality of life, investigators aim to distinguish a sensitive quantitative tool.

   Methods Interviewers who passed CITI will be trained in conducting the questionnaires to assess patients' quality of life and utility values. A set guidelines will be taught to prevent inter-examiner variability.

   Participants and target sample size 200 symptomatic patients will be recruited for this study from the dry eye clinic in SNEC. 100 patients from dry eye clinic in SNEC will be assessed with SPEED and utility assessment, and another 100 patients from dry eye clinic in SNEC will be assessed with SANDE and utility assessment.

   Visit schedules Basic eye assessments and interviewer-assisted questionnaires will be done on the same day. There will be no repeat visits required.

   Duration of study:

   One year

   Procedures:

   Assessment of Dry Eye Symptoms Basic biodata such as age, race, gender be recorded.

   • Tear break up time (TBUT) A drop of normal saline will be instilled on a fluorescein strip (Fluorets) then shaken off so that no visible drop remains. The subject is asked to look up before introduction of the fluoret into the inferior conjunctival fornix on the right then left eye.

   The participant will blink a few times and close the eyes for few seconds. The participant will then be asked to open the eyes, look ahead at the observer's forehead and not blink for as long as possible. The break up time is defined as the time between the lid opening and the first appearance of any dry spot on the cornea. The participant will be requested to close his eyes for few seconds and the procedure will be repeated for the left eye. Three reading will be taken and averaged

   Corneal fluorescein staining score Assessment of positive fluorescein staining will be assessed after recording TBUT. A scoring system will be applied as previously published by Barr et al. (Barr 1999). Briefly, there will be 5 corneal zones and 4 conjunctival regions as shown in Figure 1. The staining scale is 0-4, with 0.5 unit steps in each of the zones. The 'total' staining score will also be averaged.

   • Schirmers I test This will be done with the standard strips currently used at SERI (5 mm wide with a notch for folding) (Sno strips, Bausch & Lomb, France) without anaesthetic. The strips will be positioned over the inferior temporal half of the lower lid margin in both eyes at the same time.The study participant will be asked to close their eyes during the test. Any excessive irritation signs or reflex tearing will be noted.

   Dry eye Questionnaires Participants will be asked to score and fill up a dry eye questionnaire that assesses the symptomatic severity of dry eyes in the participant and the extent of its disruption to daily activities for the past one month.

   Two different questionnaires and utility assessment will be administered in the study;
   * SPEED Questionnaire Consist of 2 questions on frequency and severity graded on a scale of 0-3 on frequency and grade 0-4 on severity. The questionnaire allows patient to rate from 0 which is never and 3 which is all the time in frequency and 0 as no problem and 4 as intolerable in severity.
   * SANDE Questionnaire Consist of 3 questions on frequency and severity. VAS will be applied to evaluate dry eye symptoms as described by Schaumberg et al. (Schaumberg, Gulati et al. 2007). As shown in Appendix A (question 1 to 3), the scores will be recorded separately for frequency and severity of dry eye symptoms., patients will be asked to mark "X" on a 100mm line that corresponds to the degree of the symptom. A global score will be calculated by multiplying the frequency score by the severity score and taking the square root of the result (to transform back to the original scale).
   * Utility assessment Investigators will be using Time trade-off method in this study, as approved by IRB and was used in Thermal pulsation system for treatment of Meibomian Gland Dysfunction study (CRIB no: 2012/191/A). In addition, questions on socioeconomics will be administered to the patients.

   Statistics:

   Sample size calculation There will be no interim analysis. Analysis will be performed after all the subjects have completed the questionnaires or have withdrawn from the study. The distributions of the scores will be examined by histograms for normality.

   Pearson correlation coefficients (r) will be calculated between SPEED score (x) and utility value (y) for these 2 groups of patients.

   Confidence intervals will be calculated at 95% confidence level. The confidence limits are computed as;

   Expected outcomes:

   Primary Outcome
   * Difference in SPEED Questionnaire and SANDE Questionnaire that affects patient health related quality of life (HRQOL)
   * Difference in both (SPEED and SANDE) questionnaires and utility values that affects patient health related quality of life (HRQOL)

   Secondary Outcomes
   * Schirmers I reading
   * Tear break up time (TBUT)
   * Corneal fluorescein staining

   Potential problems As the 2 questionnaires used are in English and there are no validated translated questionnaires, we are limited to patients who are English-educated only. For simplicity of using validated questionnaires, we would be concentrating on English-educated patients for this study.

   Dry eye signs correlate poorly with symptoms and patient may not have an understanding of their true conditions making it more difficult to obtain accurate score. In our conservative population, sensitive questions on utility may distress the patients and therefore inability to answer the questions appropriately.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 21 years old and above and has full legal capacity to volunteer
2. Patients able to understand and complete 2 English questionnaires.
3. Symptomatic dry eye patient

Exclusion Criteria:

1. Any other specified reason as determined by clinical investigator.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from Dry Eye Clinic at Singapore National Eye Center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
• Difference in SPEED Questionnaire and SANDE Questionnaire that affects patient health related quality of life (HRQOL) | 1 day
• Difference in both (SPEED and SANDE) questionnaires and utility values that affects patient health related quality of life (HRQOL) | 1 day

SECONDARY OUTCOMES:
Production of Tear flow | 1 day
Tear break up time (TBUT) | 1 day
Corneal flourescein staining | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, PhD, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore, Singapore